CLINICAL TRIAL: NCT02557620
Title: A Randomised, Double-blind, Placebo Controlled, Double Dummy, Single-centre Trial in Healthy Subjects Comparing the Steady-state Exposure of Semaglutide Administered Subcutaneously Once Daily to Semaglutide Administered Subcutaneously Once Weekly
Brief Title: Comparing Semaglutide Administered Subcutaneously Once Daily to Semaglutide Administered Subcutaneously Once Weekly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-4215; 2014-005171-84 (EudraCT Number); U1111-1164-2741 (Other: WHO)
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- semaglutide OD + placebo semaglutide OW (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo
- placebo semaglutide OW + placebo semaglutide OD (Placebo Comparator)
  Interventions: Drug: placebo
- semaglutide OW + placebo semaglutide OD (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Administered subcutaneously (s.c., under the skin)once daily or once weekly.
  Arms: semaglutide OD + placebo semaglutide OW; semaglutide OW + placebo semaglutide OD
Drug: placebo — Administered subcutaneously (s.c., under the skin)once daily or once weekly.

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the steady-state exposure of semaglutide administered subcutaneously once daily to semaglutide administered subcutaneously once weekly in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-55 years (both inclusive) at the time of signing informed consent
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, ECG and clinical laboratory tests performed during the screeningvisit, as judged by the investigator
* Body mass index (BMI) between 20.0 and 29.9 kg/m^2 (both inclusive)
* HbA1c (glycosylated haemoglobin) below 6.5%

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive method throughout the trial including the 5 weeks follow-up period (adequate contraceptive measures as required by local regulation or practice)
* Any disorder which in the investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol
* History of pancreatitis (acute or chronic)
* Screening calcitonin equal or above 50 ng/L
* Family or personal history of Multiple Endocrine Neoplasia Type 2 (MEN2) or Medullary Thyroid Carcinoma (MTC)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Area under the semaglutide concentration-time curves | At steady-state from 0 to168 hours after dosing on day 78

SECONDARY OUTCOMES:
Maximum observed semaglutide plasma concentration | At steady-state derived from the concentration-time curves, within 168 hours from day 78
Number of treatment emergent adverse events (TEAEs) | From baseline (day 1, post-dose) to last follow-up visit (day 120)
Area under the the single dose concentration-time curve | From 0 to 300 min after administration of paracetamol (1.5 g) at day 51
Area under the the single dose concentration-time curve | From 0 to 300 min after administration of paracetamol (1.5 g) at day 79

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com